CLINICAL TRIAL: NCT03079817
Title: The Effects of Yoga Based Meditation on Proprioception in Individuals With Parkinson's Disease
Brief Title: Proprioception and Meditation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Joseph Signorile, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20151138
Record Dates: First submitted 2017-03-08; First posted 2017-03-15 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Parkinson Disease; Proprioceptive Disorders; Movement Disorders
MeSH Terms: conditions — Parkinson Disease; Somatosensory Disorders; Movement Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprioceptive Drills (Active Comparator): Includes drills during which participants perform multiplestances on a pillow, a number of different cone and line drills, reaching drills, object retrieval drills and drills using balls to disturb balance.
  Interventions: Other: Proprioceptive Drills
- Yoga Meditation (Experimental): The meditation program will use simple poses during which the participant will not move and will concentrate on each of the participant's body parts and where they are in space.
  Interventions: Other: Yoga Meditation

INTERVENTIONS:
Other: Yoga Meditation — Yoga meditation using motor imagery to perceive movement patterns
  Arms: Yoga Meditation
Other: Proprioceptive Drills — Active balance and proprioception drills
  Arms: Proprioceptive Drills

SUMMARY:
In past work is has been shown that yoga can be as effective as a standard balance or Tai Chi protocol; however, there is an inability to distinguish between the mind and body contributions of yoga training. This study will compare an accepted proprioceptive training program to a meditation program which concentrates on body awareness in individuals with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* An individual must be between 40 and 90 years of age with mild to moderate Parkinson's Disease (Hoehn & Yahr stages I-III).

Exclusion Criteria:

* Participants that have been part of a formal training program that targeted lower body strength, balance or proprioception within the past six months
* Participants that have any uncontrolled nerve (except Parkinson's patients taking appropriate medication), bone or joint, or heart disease;
* Participants that have been advised by a doctor to not exercise;
* Participants that have regularly practiced yoga at least twice per week within the past six months;
* Participants that is unable to consent;
* Participants that is a prisoner;
* Participants that are pregnant.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Joint Position Sense | 20 minutes
  The joint position sense technique for the knee involves the reduction of visual cues while moving the knee to a specific target angle, holding that target angle, returning the knee to the starting position, and then reproducing that target angle.
Tinetti balance and gait. | 3 minutes.
  A subjective evaluation of Balance and gait.

SECONDARY OUTCOMES:
8ft Up and Go | 60 seconds
  Individuals sits in a chair at the verbal cue of "go", individual rises from chair and walks as quickly as possible around a cone placed 8 ft from the front of the chair, individual returns to and sits.
Joint Kinesthesia | 20 minutes
  The Joint Kinesthesia measurement technique involves the participant sitting in the Biodex chair with visual, audio, and tactile cues reduced and the leg supported by an external movement device. The knee is placed at a predetermined angle and slowly flexed or extended at a random starting time while the participant is instructed to signal when movement is felt.
Dynamic Posturography | 5 minutes
  The participant stands on a randomly moving platform with a sonar emitter affixed to the lumbar spine. As the platform moves the linear and curvilinear displacement of the emitter is evaluated and a dynamic movement analysis core is generated.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph F Signorile, PhD, Principal Investigator — University of Miami
Locations (1):
- Laboratory of Neruomuscular Research and Active Aging, Coral Gables, Florida, United States

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886